CLINICAL TRIAL: NCT04287647
Title: Transpyloric Stenting for Refractory Gastroparesis Prior to Gastric Per-Oral Endoscopic Myotomy: a Prospective Sham Study
Brief Title: Transpyloric Stenting As a Predictor for G-POEM for Refractory Gastroparesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, A. Aziz Aadam, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00209539
Record Dates: First submitted 2019-12-04; First posted 2020-02-27 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and other care providers are blinded to whether they receive a transpyloric stent vs sham
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transpyloric stent (Active Comparator): In this group, patient's will be randomized to receive a transpyloric stent for treatment of refractory gastroparesis. They will be blinded for one month after stent placement as to whether they received a stent or sham.
  Interventions: Device: Transpyloric stent
- Sham (Sham Comparator): In this group, patient's will be randomized to sham for treatment of refractory gastroparesis. They will be blinded for one month after stent placement as to whether they received a stent or sham.
  Interventions: Other: Sham

INTERVENTIONS:
Device: Transpyloric stent — See arm/group descriptions
  Arms: Transpyloric stent
Other: Sham — Sham
  Arms: Sham

SUMMARY:
This is a prospective sham study to investigate the role of transpyloric stenting with lumen apposing metal stent (LAMS) as a predictor for clinical response to gastric per-oral endoscopic pyloromyotomy (GPOEM) for refractory gastroparesis. The study hypothesizes that clinical improvement with transpyloric stenting in patients with refractory gastroparesis is a predictor of subsequent clinical success of GPOEM.

DETAILED DESCRIPTION:
Gastroparesis is defined as a complex syndrome of symptoms including early satiety, post-prandial fullness, nausea, vomiting, bloating, and upper abdominal pain with a corresponding objective delay in gastric emptying in the absence of mechanical obstruction. Recent epidemiologic data has shown a substantial increase of 158% in hospitalizations related to gastroparesis in recent years. The pathogenesis underlying gastroparesis is complex with multiple potential underlying mechanisms including impaired gastric accommodation, autonomic neuropathy, vagal nerve injury, uncoordinated gastric contractility, and pyloric dysfunction.

Effective and durable medical treatment of gastroparesis has remained clinically challenging. Currently metoclopramide is the only medication approved by the U.S. Food and Drug Administration (FDA) for diabetic gastroparesis, and treatment courses are recommended to be limited to a maximum of 12 weeks due to the risk of the irreversible side effect of tardive dyskinesia. Surgical treatments for gastroparesis also remain limited, with sparse existing data to support the use of implanted gastric electrical stimulation for treatment of refractory gastroparesis, which is currently approved by the FDA only for compassionate use. More recently, surgical pyloroplasty has been examined in treatment of gastroparesis, which has long been recognized as a technique to improve gastric drainage for mechanical obstructions and during elective vagotomy after gastric surgery. A recent study examined surgical pyloroplasty in 28 patients with post-surgical gastroparesis with 83% patients reporting significant clinical improvement at one-month follow-up but current surgical literature remains limited in this area and has focused primarily on post-surgical gastroparesis.

Given the lack of effective treatment options, endoscopic therapies for gastroparesis have recently been investigated as adjunctive or alternative methods to treat gastroparesis. Pyloric dysfunction characterized by pyloric restriction or pylorospasm with prolonged periods of increased pyloric tone and contractions has been brought to attention as an area of targetable therapy for a subset of patients with gastroparesis. Pyloric botulinum toxin injections initially demonstrated improvement in gastric emptying after treatment, but subsequent results from double-blinded placebo-control studies failed to demonstrate a difference in symptoms compared to placebo.

Transpyloric stenting was initially reported in 2013 in three cases of refractory gastroparesis with placement of a double layered, fully-covered, Niti-S self-expandable metal stent (TaeWoong Medical) across the pylorus with improvement in gastric emptying and symptoms in all three patients. A subsequent study of 30 patients with refractory gastroparesis who underwent transpyloric stenting demonstrated high technical success of stent placement (98%) with improvement of clinical symptoms in 75% of patients and 4-hour gastric emptying studies in 69% of patients. Stent migration was found to occur in 59% of patients without any associated adverse events. Current focus on transpyloric stenting in gastroparesis centers around determining optimal stent type and method of stent anchorage as well as the role of transpyloric stenting in treatment given lack of long-term durability.

With advancements in endoscopic submucosal dissection, G-POEM has recently come in to light as a minimally invasive technique to treat refractory gastroparesis. Esophageal endoscopic myotomy has previously been well-described as a procedure for treatment of achalasia, and this technique was adopted by in 2013 with the first G-POEM for refractory gastroparesis. A subsequent multicenter study in 2017 reported on 30 patients with refractory gastroparesis who underwent G-POEM with a technical success rate of 100%. At 5.5-month follow-up, 86% of patients were found to have clinical response. Repeat gastric emptying studies after G-POEM also normalized or improved in 47% and 37% of patients respectively. G-POEM has now gained both national and international recognition in succeeding studies as a feasible and safe technique to effectively treat refractory gastroparesis in a subset of patients.

Identifying predictors of success of G-POEM for treatment of gastroparesis is essential in further recognizing appropriate patients who would benefit from this therapy. As transpyloric stenting and G-POEM share underlying mechanisms of disruption of the pylorus, the investigators propose that improvement with transpyloric stenting in patients with refractory gastroparesis can be a predictor of subsequent response with G-POEM.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than 18 years of age with gastroparesis refractory to standard medical therapy (lifestyle and diet modifications, prokinetics) or contraindication to standard therapies (e.g. allergies to prokinetic agents)
* Patients with diabetic, idiopathic or post-surgical gastroparesis
* Patients with confirmed diagnosis of gastroparesis via gastric emptying study (abnormal gastric emptying will be defined as ≥10 % residual activity at 4 h on a standardized nuclear medicine TC-99 m sulfur colloid solid-phase gastric emptying study)

Exclusion Criteria:

* Patients with prior history of gastroenteric anastomosis or any GI surgeries with pyloric involvement
* Patients with gastroesophageal malignancy
* Patients who are unable to tolerate upper endoscopy secondary to cardiopulmonary instability or other contraindications to endoscopy
* Patients with cirrhosis
* Patients who are pregnant or breastfeeding
* Patients with uncorrectable coagulopathy defined by INR >1.5 or platelets <50

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Clinical response will be assessed by the gastroparesis cardinal symptom index (GCSI) scores | 1-2 years
  GCSI assessment is based off an average of 16 questions that are scored from 0-5, with higher scores indicating a worse clinical outcome.

SECONDARY OUTCOMES:
Age | 1-2 years
  Assessed in years
Weight | 1-2 years
  Assessed in kilograms
Height | 1-2 years
  Assessed in inches
BMI | 1-2 years
  Assessed in kg/m^2
Adverse events | 1-2 years
  Assessed based on current American Society for Gastrointestinal Endoscopy (ASGE) guideline definitions for endoscopic adverse events
Procedure length | intraoperative
  Assessed in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No